CLINICAL TRIAL: NCT00201786
Title: Phase II Trial of Pentostatin in Steroid Refractory Acute Graft Versus Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Craig Hofmeister, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0301
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Graft-Versus-Host Disease
Keywords: Corticosteroids
MeSH Terms: conditions — Graft vs Host Disease | interventions — Pentostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pentostatin (Experimental): Pentostatin is given at a dose of 1.5 mg/m2/day IV x 3 consecutive days. Each IV infusion of pentostatin will be administered over 20-30 minutes in 100-250 ml of D5W or NS.
  Interventions: Drug: Pentostatin

INTERVENTIONS:
Drug: Pentostatin — Pentostatin is given at a dose of 1.5 mg/m2/day IV x 3 consecutive days. Each IV infusion of pentostatin will be administered over 20-30 minutes in 100-250 ml of D5W or NS. To prevent nephrotoxicity, patients will also receive 500 ml normal saline as pre- and post drug hydration (total 1000 ml).
  Other Names: (Nipent®, Supergen)

SUMMARY:
This study will evaluate the response rate to treatment with pentostatin in steroid-refractory acute graft versus host disease.

ELIGIBILITY:
Inclusion Criteria:

* Must have biopsy proven grade II-IV acute GVHD refractory to systemic corticosteroids
* No chronic GVHD
* Age ≥ 18 years
* Evidence of myeloid engraftment (ANC ≥ 0.5 x 109/l)
* Performance status 0-3

Exclusion Criteria:

* Patients on mechanical ventilation or who have resting O2 saturation <90% by pulse-oximetry.
* Patients on renal dialysis or who have an estimated creatinine clearance of < 30 ml/min/1.73 m2.
* Patients with documented clinical infection (progressive symptoms despite antibiotics or continued fever) cannot be enrolled on study until infection is controlled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-07; Primary Completion 2007-10 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the response rate (complete and partial) to treatment with pentostatin in steroid-refractory acute GVHD (graft-versus-host disease). | up to 2 years

SECONDARY OUTCOMES:
Investigate the pharmacokinetics of pentostatin in patients with acute GVHD to correlate the response with area under the curve (AUC). | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hofmeister, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Result] Poi MJ, Hofmeister CC, Johnston JS, Edwards RB, Jansak BS, Lucas DM, Farag SS, Dalton JT, Devine SM, Grever MR, Phelps MA. Standard pentostatin dose reductions in renal insufficiency are not adequate: selected patients with steroid-refractory acute graft-versus-host disease. Clin Pharmacokinet. 2013 Aug;52(8):705-12. doi: 10.1007/s40262-013-0064-7. PMID 23588536
- See also: Jamesline — http://cancer.osu.edu